CLINICAL TRIAL: NCT02110069
Title: A Randomized Phase 2 Study of Vincristine Versus Sirolimus to Treat High Risk Kaposiform Hemangioendothelioma (KHE).
Brief Title: A Study to Compare Vincristine to Sirolimus for Treatment of High Risk Vascular Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was challenged by the incidence of KHE with KMP as this continued to be extremely rare, and very sporadic. In July of 2019 grant renewal funding ended.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Denise Martin Adams, Associate Professor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIR-DA-1202; 1R01FD004363-01A1 (FDA); 2013-2339 (Other: CCHMC IRB)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Kaposiform Hemangioendothelioma (KHE); Kasabach-Merritt Syndrome; Tufted Angioma
Keywords: KHE; Vascular anomaly; Kasabach-Merritt Syndrome; Tufted angioma; hemangioendothelioma
MeSH Terms: conditions — Kaposiform Hemangioendothelioma; Kasabach-Merritt Syndrome; Tufted angioma; Vascular Malformations; Hemangioendothelioma | interventions — Vincristine; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vincristine (Active Comparator): Induction phase: participants assigned to vincristine will receive vincristine weekly at a dose of 0.05mg/kg/dose IV (for participants less than 10kg) or a dose of 1.5 mg/m2/dose (for participants greater than 10kg) for 2 months.
  Maintenance: if participants continue to receive vincristine weekly for 2 months, every 2 weeks for 5 months and every 3 weeks for 5 months.
  Interventions: Drug: Vincristine
- Sirolimus (Experimental): Sirolimus will be administered at a dose of 0.8mg/m2/dose twice a day on a continuous dosing schedule throughout the trial for participants randomized to Sirolimus or for participants who fail vincristine may cross-over to the sirolimus arm.
  Sirolimus trough levels will be maintained between 10-15 ng/ml.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Vincristine — Vincristine dose dependent upon weight. Weekly for 2 months (Induction); Weekly 2 months; every 2 weeks for next 5 months; every 3 weeks for 5 months (Maintenance)
  Other Names: Oncovin; Vincasar® PFS; Vincrex
  Arms: Vincristine
Drug: Sirolimus — Continuous dosing to maintain trough level of 10-15ng/ml.
  Other Names: Rapamune
  Arms: Sirolimus

SUMMARY:
In this research study we want to learn more about which treatment works better for patients diagnosed with a vascular tumor called Kaposiform Hemangioendothelioma (KHE) or other high risk vascular tumors such as Tufted Angioma (TA). In these tumors, the blood cells that help your blood clot called platelets become trapped in the tumor causing swelling, pain, and bruising. Vascular tumors can be life threatening. There are few medical treatments that will work to shrink the vascular tumor. Some doctors will use steroids and vincristine to try and shrink vascular tumors.

In this research study, the study doctor will compare two different drugs to see which one will work better to help shrink your vascular tumor. One of the drugs is vincristine. Vincristine is approved by the Food and Drug Administration (FDA) to treat people with cancer. Vincristine is used to stop the abnormal cells from growing such as cells that make up blood vessels.

The other drug to be used in this study is sirolimus. Sirolimus is currently approved by the Food and Drug Administration (FDA) to prevent transplanted organ rejection. Sirolimus is not approved by the FDA for treatment of vascular abnormalities and is considered experimental. Sirolimus belongs to a class of drugs call 'mTOR inhibitors'. mTOR (mammilian target of rapamycin) helps cells to grow and may also help blood vessels to grow in a more normal fashion. Sirolimus is currently being tested in patients with vascular tumors and cancer. In vascular tumors, we hope sirolimus will stop the blood vessel growth.

Funding Source: FDA - OOPD (Office of Orphan Products Development)

DETAILED DESCRIPTION:
Kaposiform hemangioendotheliomas (KHE) are extremely rare life threatening tumors which can be associated with Kasabach-Merritt Phenomenon consisting of profound thrombocytopenia and hypofibrinogenemia causing a significant risk of bleeding and an associated mortality rate as high as 20% to 30%. Despite the severity of potential complications, we lack uniform guidelines for the treatment and response to treatment of children and young adults with these tumors. KHE patients have been treated with a multitude of aggressive drug regimens without prospective evaluation of response or safety. Presently, vincristine is considered the standard of practice. We have treated a subset of these patients on study SIR-DA-0901 (FDA Grant# 5RO1FD003712-01). This study is a phase II trial assessing the efficacy and safety of sirolimus for the treatment of complicated vascular anomalies. Although the numbers are small, the response has been extremely promising with excellent tolerability. There is pre-clinical and clinical data supporting the essential regulatory function of the PI3 kinase/AKT/mTOR pathway in vascular growth and organization which suggests a therapeutic target for patients with complicated vascular anomalies. The overall goal of this trial is to objectively assess the efficacy of sirolimus compared to vincristine for the treatment of patients with high risk KHE.

Hypothesis: Sirolimus treatment for children and young adults with Kaposiform hemangioendotheliomas will be more effective than vincristine, assessed by time to response in an induction period and provide equivalent safety parameters.

Study Rationale We propose a multi-center, phase II trial with participation from 8 sites. The study will consist of two phases. The first of these is an initial induction phase in which vincristine and steroids will be compared to sirolimus and steroids. Response in the induction phase will be assessed as time to hematologic response. At the end of induction phase, cross over can occur if there is failure to respond. Part 2 is a maintenance phase which will be 1 year in length. Continued safety and efficacy data will be collected during maintenance and there will be cross over at any time for patients who lose their response following induction. Failure will be defined as worsening of hematological parameters on two separate laboratory evaluations at any time during maintenance or if they meet the definition of progressive disease following response assessments. Formal response in maintenance will be evaluated by imaging studies, functional assessment, and quality of life as per study SIR-DA-0901. Present therapies are very limited and new therapies are desperately needed for this devastating disease. Based on our preliminary data, there is a very good rationale for sirolimus therapy in KHE patients and so a phase II trial is urgently needed to determine if this therapy is to become the new standard of care for KHE patients.

Our secondary aims will be addressing biomarker analysis. There are limited studies describing the biology of these tumors. Per study SIR-DA-0901 there is some preliminary data indicating the importance of VEGF-C and other upregulated markers in the mTor pathway. This needs to be further investigated especially in KHE patients. Furthermore there are no clear objective measurements to determine response data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: All patients must have one of the following vascular anomalies as determined by clinical, radiologic and histologic criteria (when possible). Biopsy strongly recommended (but not required) with suggested immunostains: CD34, PROX-1 or D240, Glut-1 and MIB-1.

  1. Kaposiform Hemangioendotheliomas
  2. Tufted angioma

High Risk Stratification: In addition to the above diagnosis, all of the following criteria need to be met:

a. Kasabach Merritt Syndrome defined at a platelet counts less than 50,000 K/µl and/or fibrinogen level < 100 mg/dl at the time of diagnosis.

* Age: Patients must be 0 - 31 years of age at the time of study entry. Enrollment includes patients of both genders and all ethnic groups.
* Organ function requirements:

  1. Adequate liver function defined as:

     1. Total bilirubin ≤ 1.5 x ULN for age, and
     2. SGPT (ALT) ≤ 5 x ULN for age, and
     3. Serum albumin >/= 2 g/dL.
     4. Fasting LDL cholesterol of <160 mg/dL
     5. Fasting triglyceride <400 mg/dl
  2. Adequate Bone Marrow Function defined as:

     1. Peripheral absolute neutrophil count (ANC) >/= 1000/uL
     2. Hemoglobin >/= 8.0 g/dL (may receive RBC transfusions)
     3. No Platelet requirement
  3. Adequate Renal Function Defined as:

     1. A serum creatinine based on age as follows:

        Age (Years) Maximum Serum Creatinine (mg/dL)
        * 5 0.8 6 to ≤10 1.0 11 to ≤15 1.2 >15 1.5
     2. Urine protein to creatinine ratio (UPC) < 0.3 g/l
* Performance Status: Karnofsky >/= 50 (≥16 years of age) and Lansky >/= 50 for patients <16 years of age.
* Prior therapy

  1. Patients who have undergone surgical resection or interventional radiology procedures for disease control are eligible if they meet all inclusion criteria after surgery/procedure
  2. Surgery: At least 2 weeks since undergoing any major surgery
  3. Radiation: > 6 months from involved field radiation
  4. Prior vincristine therapy is permitted. Patients may also have received up to 2 doses of vincristine prior to randomization.

Exclusion Criteria:

* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration).
* Patients who require medications that are strong inhibitors/inducers CYP3A4 enzyme activity, including anticonvulsants, (Appendix II) to control concurrent medical conditions are not eligible. Patients who discontinue use of prohibited medications with a one week washout prior to start of study treatment are eligible.
* Known history of HIV seropositivity or known immunodeficiency. Testing is not required unless a condition is suspected.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of sirolimus (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection). A gastric tube or nasogastric tube is allowed.
* Females who are pregnant or breast feeding.
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during the period they are receiving the study drug and for 3 months thereafter. Abstinence is an acceptable method of birth control. Females of childbearing potential will be given a pregnancy test within 7 days prior to administration of study treatment and must have a negative urine or serum pregnancy test.
* Patients who have received prior treatment with an mTOR inhibitor.
* Patients unwilling or unable to comply with the protocol or who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Patients who currently have an uncontrolled infection, defined as receiving intravenous antibiotics.

Max Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Adams, MD, Principal Investigator — Boston Children's Hospital
Locations (7):
- United States (7):
  - Lucille Packard Children's Hospital Stanford, Palo Alto, California
  - Emory Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cincinnati Children's Hospital Medical Center Hemangioma and Vascular Malformation Center — http://www.cincinnatichildrens.org/service/h/hemangioma/default/
- See also: National Organization of Vascular Anomalies — http://www.novanews.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Vincristine: Induction phase: participants assigned to vincristine will receive vincristine weekly at a dose of 0.05mg/kg/dose IV (for participants less than 10kg) or a dose of 1.5 mg/m2/dose (for participants greater than 10kg) for 2 months.
  Maintenance: if participants continue to receive vincristine weekly for 2 months, every 2 weeks for 5 months and every 3 weeks for 5 months.
  Vincristine: Vincristine dose dependent upon weight. Weekly for 2 months (Induction); Weekly 2 months; every 2 weeks for next 5 months; every 3 weeks for 5 months (Maintenance)
- Sirolimus: Sirolimus will be administered at a dose of 0.8mg/m2/dose twice a day on a continuous dosing schedule throughout the trial for participants randomized to Sirolimus or for participants who fail vincristine may cross-over to the sirolimus arm.
  Sirolimus trough levels will be maintained between 10-15 ng/ml.
  Sirolimus: Continuous dosing to maintain trough level of 10-15ng/ml.
Period: Overall Study
Arm/Group | Vincristine | Sirolimus
Started | 2 | 2
Completed (second subject came off study at maintenance course 6 as family moved out of the country) | 0 (subject was switched to sirolimus at maintenance course 7 for failure on Vincristine) | 2 (1 subject was takend off protocol treatment at 10 months of maintenance for disease response.)
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: no analysis was performed as study was closed early
Groups:
- Total: Total of all reporting groups
Arm/Group | Vincristine | Sirolimus | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: There was no analysis as study was closed early
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Number of participants with platelet count & fibrinogen levels [Number; unit: participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Hematologic Parameters
Description: Hematologic parameters are defined as a platelet count greater than 100,000/uL (or a 2 times increase in platelet count compared to baseline) and a fibrinogen level greater than 150mg/dl.
Time Frame: 2 months
Population: no analysis was performed due to study being closed for low enrollment
Arm/Group | Vincristine | Sirolimus
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Serious and Non-Serious Adverse Events
Description: Serious and non-serious adverse events will be recorded for all participants and graded using CTCAE v4.0 (Common Toxicity Criteria for Adverse Effects). Adverse event rates will be calculated for both sirolimus and vincristine.
Time Frame: 2 months; 12 months
Population: study was closed early due to slow enrollment
Arm/Group | Vincristine | Sirolimus
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Evaluation of Disease Response - Maintenance
Description: Disease evaluation will be measured using a combination of quality of life assessments, clinical parameters, and radiologic images.
Time Frame: 6 months; 12 months
Population: no analysis was performed
Arm/Group | Vincristine | Sirolimus
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Serious and Non Serious Adverse Events - Maintenance
Description: Serious adverse events and adverse events will be graded according to CTCAE v4.0. Adverse event rates will be calculated for both sirolimus and vincristine.
Time Frame: 6 months; 12 months
Population: no data analyzed as study was closed early
Arm/Group | Vincristine | Sirolimus
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in the Serum Levels of KHE Biomarkers
Description: The following KHE biomarkers will be evaluated vascular endothelial growth factor A, C, and D (VEGF-A, C, D_, IL-8 (interleukin), Pleiotrophin, IGF-1 (insulin-like growth factor), endothelin-1, thrombospondin and angiopoietin 1 and 2.
Time Frame: Baseline, 2 months, 6 months, and 12 months
Population: no analysis performed as study was closed early
Arm/Group | Vincristine | Sirolimus
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Identify Genetic Variants in Drug Metabolism Enzymes.
Description: Single nucleotide polymorphism array analysis to obtain genetic information on variants in drug metabolism enzymes that affect sirolimus and vincristine metabolism.
Time Frame: Baseline
Population: study closed early due to slow enrollment
Arm/Group | Vincristine | Sirolimus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 months for 2 subjects 12 months for 1 subject 6 months for 1 subject
Arm/Group | Vincristine | Sirolimus
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vincristine (N=2) | Sirolimus (N=2)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) — Subject admitted to hospital and test positive for adenovirus
Lung infection (Infections and infestations) | 1 (1) | 0 (0) — Subject tested positive for RSV
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — Central Line Associated BloodStream Infection
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vincristine (N=2) | Sirolimus (N=2)
Fever (Infections and infestations) | 1 (1) | 1 (1) — Grade 2
anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Grade 2
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT02110069/Prot_SAP_000.pdf